CLINICAL TRIAL: NCT05737940
Title: A Phase IIb Randomised, Double-blind, Placebo-controlled, Multi-centre, Dose-ranging Study of AZD3427 in Participants With Heart Failure and Pulmonary Hypertension Due to Left Heart Disease (WHO Group 2)
Brief Title: A Study of AZD3427 in Participants With Heart Failure and Pulmonary Hypertension Group 2
Acronym: Re-PHIRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D8330C00003
Record Dates: First submitted 2023-01-20; First posted 2023-02-21 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Hypertension (World Health Organization Group 2); Heart Failure
Keywords: Pulmonary Hypertension; Heart Failure; Left Heart Disease; WHO Group 2; Dose-ranging Study; Pulmonary vascular resistance
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AZD3427 Dose A (Experimental): The participants will receive single dose of AZD3427 Dose A every 2 weeks for 24 weeks from Day 1 to Day 155.
  Interventions: Drug: AZD3427
- AZD3427 Dose B (Experimental): The participants will receive single dose of AZD3427 Dose B every 2 weeks for 24 weeks from Day 1 to Day 155.
  Interventions: Drug: AZD3427
- AZD3427 Dose C (Experimental): The participants will receive single dose of AZD3427 Dose C every 2 weeks for 24 weeks from Day 1 to Day 155.
  Interventions: Drug: AZD3427
- Placebo (Placebo Comparator): The participants will receive single dose of placebo every 2 weeks for 24 weeks from Day 1 to Day 155.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD3427 — The participants will receive AZD3427 SC injection single dose of either Dose A or Dose B or Dose C every 2 weeks for 24 weeks.
  Arms: AZD3427 Dose A; AZD3427 Dose B; AZD3427 Dose C
Drug: Placebo — The participants will receive SC injection of placebo single dose every 2 weeks for 24 weeks.
  Arms: Placebo

SUMMARY:
This study is intended to assess the ability of AZD3427 to reduce pulmonary vascular resistance (PVR) after 24 weeks of treatment in participants with heart failure (HF) and pulmonary hypertension (PH) Group 2

DETAILED DESCRIPTION:
This study is a randomized, placebo-controlled, multi-centre, dose-ranging study of AZD3427 in participants with heart failure and pulmonary hypertension due to left heart disease (World Health Organisation [WHO] Group 2).

Approximately 220 participants will be randomised to 4 treatment groups (in a 1:1:1:1 ratio) to receive a subcutaneous (SC) injection of AZD3427 or placebo every 2 weeks for 24 weeks.

This study will evaluate 3 dose levels of AZD3427: Dose A, Dose B, and Dose C. Dose modification is not applicable for this study.

The study will be conducted in approximately 60 study centres across an estimated 15 countries.

The study will include approximately 16 study visits: 2 visits during the Screening Period,13 visits during the Treatment Period, and one visit during the Follow-up Period.

The expected total duration of the study is 32 to 37 weeks, depending on the length of the Screening Period.

ELIGIBILITY:
Inclusion criteria:

1. Participant must be ≥ 18 years of age inclusive.
2. Participants must have a pre-existing diagnosis of HF, NYHA function class (FC) II to IV, and a pre-existing diagnosis of PH-LHD or likely or intermediate probability of Pulmonary hypertension due to left heart disease (PH-LHD) as per 2022 Pulmonary hypertension due to left heart disease European Society of Cardiology/European Respiratory Society (ESC/ERS) guidelines. Participants must be on stable HF standard of care medication, including diuretics.
3. Participants must have a combination of echocardiographic parameters that show intermediate or high probability of PH as per 2022 ESC/ERS guidelines.
4. Participants must have an on-study elevated pulmonary artery pressure from RHC performed as per RHC manual provided by the Sponsor, at Screening Visit 2:

   1. PAWP ≥ 15 mmHg
   2. mPAP ≥ 20 mmHg
5. Minimum body weight of 45 kg (inclusive).
6. Capable and willing of giving signed informed consent.

Exclusion Criteria

1. Diagnosis of PH in World Health Organization (WHO) Group 1, WHO Group 3, WHO Group 4, or WHO Group 5.
2. Historical or current evidence of a clinically significant disease or disorder.
3. Decompensated HF or hospitalisation due to decompensated HF.
4. Any contraindications to RHC.
5. History of hypersensitivity to SC injections or devices.
6. History of hypersensitivity to drugs with a similar chemical structure or class to AZD3427 or any component of AZD3427 drug product, or ongoing clinically important allergy/hypersensitivity.
7. Known lung disease with Forced expiratory volume in the first second (FEV1) < 30% of predicted.
8. Congenital long QT syndrome.
9. Cardiac ventricular arrhythmia which requires treatment. Participants with atrial fibrillation or flutter and controlled ventricular rate are permitted.
10. History of or anticipated heart transplant or ventricular assist device implantation.
11. Any known planned (scheduled) highly invasive Cardiovascular (CV) procedure (eg, coronary revascularisation, ablation of atrial fibrillation/flutter, valve repair/replacement, aortic aneurysm surgery, etc).
12. Participants who have previously received AZD3427.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Pulmonary Vascular Resistance (PVR) | Baseline to Week 25
  To evaluate the effect of AZD3427 on PVR parameter compared with placebo as measured by right heart catheterization (RHC) after 24 weeks of treatment in participants with HF and PH Group 2.

SECONDARY OUTCOMES:
Change from baseline in Mean pulmonary arterial pressure (mPAP) | Baseline to Week 25
  To evaluate the effect of AZD3427 compared with placebo on mPAP parameter after 24 weeks of treatment in participants with HF and PH Group 2.
Change from baseline in Pulmonary artery wedge pressure (PAWP) | Baseline to Week 25
  To evaluate the effect of AZD3427 compared with placebo on PAWP parameter after 24 weeks of treatment in participants with HF and PH Group 2.
Change from baseline in cardiac output | Baseline to Week 25
  To evaluate the effect of AZD3427 compared with placebo on cardiac output parameter after 24 weeks of treatment in participants with HF and PH Group 2.
Change from baseline in Stroke Volume (SV) | Baseline to Week 25
  To evaluate the effect of AZD3427 compared with placebo on SV parameter after 24 weeks of treatment in participants with HF and PH Group 2.
Change from baseline in Ejection fraction (EF) | Baseline to Week 25
  To evaluate the effect of AZD3427 compared with placebo on EF parameter after 24 weeks of treatment in participants with HF and PH Group 2.
Change from baseline in left ventricular global longitudinal strain (LVGLS) | Baseline to Week 25
  To evaluate the effect of AZD3427 compared with placebo on LVGLS parameter after 24 weeks of treatment in participants with HF and PH Group 2.
Change from baseline in pulmonary arterial systolic pressure (PASP) | Baseline to Week 25
  To evaluate the effect of AZD3427 compared with placebo on PASP parameter after 24 weeks of treatment in participants with HF and PH Group 2.
Change from baseline in right ventricle/left ventricle (RV/LV) ratio | Baseline to Week 25
  To evaluate the effect of AZD3427 compared with placebo on RV/LV parameter after 24 weeks of treatment in participants with HF and PH Group 2.
Change from baseline in right ventricular outflow tract acceleration time (RVOT AT) | Baseline to Week 25
  To evaluate the effect of AZD3427 compared with placebo on RVOT AT parameter after 24 weeks of treatment in participants with HF and PH Group 2.
Change from baseline in Tricuspid regurgitation velocity (TRV) | Baseline to Week 25
  To evaluate the effect of AZD3427 compared with placebo on TRV parameter after 24 weeks of treatment in participants with HF and PH Group 2.
Change from baseline in TAPSE/PASP [Tricuspid annular plane systolic excursion/ Pulmonary arterial systolic pressure] | Baseline to Week 25
  To evaluate the effect of AZD3427 compared with placebo on TAPSE/PASP parameter after 24 weeks of treatment in participants with HF and PH Group 2.
Change from baseline in systemic vascular resistance | Baseline to Week 25
  To evaluate the effect of AZD3427 compared with placebo on systemic vascular resistance parameter after 24 weeks of treatment in participants with HF and PH Group 2.
Change from baseline in 6-minute walking distance (6MWD) | Baseline to Week 25
  To evaluate the effect of AZD3427 compared with placebo on function and symptoms using 6MWD parameter after 24 weeks of treatment in participants with HF and PH Group 2.
Change from baseline in Kansas City Cardiomyopathy Questionnaire total symptom score (KCCQ TSS) | Baseline to Week 25
  To evaluate the effect of AZD3427 compared with placebo on function and symptoms using KCCQ TSS parameter after 24 weeks of treatment in participants with HF and PH Group 2. The score ranges from 0 to 100, where a higher score represents a better patient outcome.
Change from baseline in New York Heart Association Functional Class (NYHA FC) | Baseline to Week 25
  To evaluate the effect of AZD3427 compared with placebo on function and symptoms using NYHA FC parameter after 24 weeks of treatment in participants with HF and PH Group 2.
Change from baseline in serum creatinine | Baseline to Week 13 and Week 25
  To evaluate the effect of AZD3427 compared with placebo using serum creatinine parameter after 12 and 24 weeks of treatment in participants with HF and PH Group 2.
Change from baseline in N-terminal prohormone of brain natriuretic peptide (NT-proBNP) | Baseline to Week 13 and Week 25
  To evaluate the effect of AZD3427 compared with placebo using NT-proBNP parameter after 12 and 24 weeks of treatment in participants with HF and PH Group 2.
Change from baseline in cystatin C | Baseline to Week 13 and Week 25
  To evaluate the effect of AZD3427 compared with placebo using cystatin C parameter after 12 and 24 weeks of treatment in participants with HF and PH Group 2.
Change from baseline in eGFR (estimated glomerular filtration rate) | Baseline to Week 13 and Week 25
  To evaluate the effect of AZD3427 compared with placebo using eGFR parameter after 12 and 24 weeks of treatment in participants with HF and PH Group 2.
Pharmacokinetics (AZD3427 serum exposure) | On Day 15, Day 29, Day 85, Day 127, Day 169, and Day 211
  Serum concentration of AZD3427 summarised by timepoints and dose level.
Number of participants with presence of Anti-drug antibodies (ADAs) | On Day 1, Day 15, Day 29, Day 85, Day 169, and Day 211
  To evaluate the immunogenicity of AZD3427 using ADA parameter.
Evaluation of positive ADA titer | On Day 1, Day 15, Day 29, Day 85, Day 169, and Day 211
  To evaluate the immunogenicity of AZD3427 as measured by ADAs.

OTHER OUTCOMES:
Number of participants with adverse events and serious adverse events | From Randomization (Day 1) up to Follow-up Visit (Day 211)
  To evaluate the safety and tolerability of AZD3427 as compared to placebo in participants with HF and PH Group 2

CONTACTS AND LOCATIONS:
Locations (56):
- United States (7):
  - Research Site, Beverly Hills, California
  - Research Site, La Jolla, California
  - Research Site, New Haven, Connecticut
  - Research Site, Baltimore, Maryland
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Rock Hill, South Carolina
- Austria (2):
  - Research Site, Linz
  - Research Site, Vienna
- Canada (7):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (4):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Guangzhou
  - Research Site, Kunming
- Research Site, Prague, Czechia
- Denmark (2):
  - Research Site, Aarhus
  - Research Site, Copenhagen
- Germany (4):
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Frankfurt
  - Research Site, Jena
- Italy (5):
  - Research Site, Brescia
  - Research Site, Genoa
  - Research Site, Marche
  - Research Site, Milan
  - Research Site, Trieste
- Japan (7):
  - Research Site, Bunkyō City
  - Research Site, Kasugai-shi
  - Research Site, Kure-shi
  - Research Site, Nagoya
  - Research Site, Sapporo
  - Research Site, Sunto-gun
  - Research Site, Toyama
- Netherlands (3):
  - Research Site, Deventer
  - Research Site, Heerlen
  - Research Site, Tilburg
- Poland (5):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Spain (4):
  - Research Site, Majadahonda
  - Research Site, Seville
  - Research Site, Toledo
  - Research Site, Valencia
- Sweden (2):
  - Research Site, Gothenburg
  - Research Site, Huddinge
- United Kingdom (3):
  - Research Site, Cambridge
  - Research Site, Clydebank
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/